CLINICAL TRIAL: NCT06216561
Title: A Phase I Trial of Intraperitoneal LSTA1 in Patients Undergoing Cytoreductive Surgery and HIPEC for Peritoneal Surface Malignancy
Brief Title: Intraperitoneal LSTA1 in CRS-HIPEC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: closed early due to low (0) accrual
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Joel Baumgartner, Associate Professor of Surgery, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSD 807804
Record Dates: First submitted 2023-12-22; First posted 2024-01-22 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer; Ovarian Carcinoma; Appendix Cancer; Peritoneal Metastases
MeSH Terms: conditions — Colorectal Neoplasms; Ovarian Neoplasms; Appendiceal Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Intervention Model Description: Unblinded, randomized 2:1 to CRS-HIPEC + LSTA1 vs. CRS-HIPEC alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CRS-HIPEC + LSTA1 (Experimental): Experimental Arm
  Interventions: Drug: CRS-HIPEC + LSTA1
- CRS-HIPEC alone (Active Comparator): Control Arm
  Interventions: Procedure: CRS-HIPEC alone

INTERVENTIONS:
Drug: CRS-HIPEC + LSTA1 — LSTA1 given with hyperthermic intraperitoneal chemotherapy (HIPEC) at time of cytoreductive surgery (CRS)
  Other Names: Cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC) + Advanced Solid TumorsCertepetide (LSTA1)
  Arms: CRS-HIPEC + LSTA1
Procedure: CRS-HIPEC alone — Hyperthermic intraperitoneal chemotherapy (HIPEC) alone (without LSTA1) at time of cytoreductive surgery (CRS)
  Arms: CRS-HIPEC alone

SUMMARY:
This Study is designed to test an investigational product (IP) called LSTA1 (Study drug). LSTA1 is a drug designed to improve the delivery of anti-cancer treatments, such as chemotherapy. Improved delivery of chemotherapy may result in improved anti-cancer effects when given with hyperthermic intraperitoneal chemotherapy (HIPEC) in patients with peritoneal metastases. Participants will be randomized to receive LSTA1 with HIPEC or HIPEC alone (without LSTA1) at the time of surgery.

DETAILED DESCRIPTION:
Given the high recurrence and disease-related mortality in patients with peritoneal metastases from appendiceal, colorectal, and ovarian cancer after cytoreductive surgery and hyperthermic intraperitoneal chemotherapy (CRS-HIPEC), use of an agent to improve operative tumor delivery of co-administered anticancer drugs during HIPEC would potentially have significant impact on oncologic outcomes.

Safety of LSTA1 has been demonstrated in the context of metastatic pancreatic cancer when administered intravenously with cytotoxic chemotherapy, but the investigators wish to determine its safety and potential efficacy when administered intraperitoneally with HIPEC in patients with peritoneal metastases from appendiceal, colorectal, and ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Participants must have histologically confirmed non-mucinous (< 50% mucin) colorectal, ovarian, or appendiceal carcinoma with peritoneal metastases who are candidates for (cytoreductive surgery and CRS-HIPEC and have at least one peritoneal tumor nodule > 5 mm (as determined by routine preoperative imaging and confirmed by intraoperative assessment).
4. Eligible and intended to undergo CRS-HIPEC per the investigators. This includes assessment of axial imaging (computed tomography, magnetic resonance imaging, positron emission tomography scan) of chest, abdomen, and pelvis, within 30 days of screening, which reveals peritoneal metastases amenable to complete cytoreduction per the investigators (i.e. limited small bowel/mesenteric metastases), lack of extra-peritoneal metastases (including intra-hepatic and pulmonary metastases), and lack of untreated biliary, gastrointestinal, and urologic obstruction.
5. Age ≥ 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status < 2.
7. Women of child-bearing potential with negative pregnancy test prior to undergoing CRS-HIPEC.
8. Adequate contraception for participants able to cause a pregnancy:

Exclusion Criteria:

1. Participants who do not receive HIPEC at the time of CRS.
2. Any major surgery or irradiation within 30 days prior to prior to planned date of CRS-HIPEC.
3. Active infection (viral, fungal, or bacterial) requiring systemic therapy.
4. Known active hepatitis B virus (HBV), hepatitis C virus (HCV), tuberculosis, or human immunodeficiency virus (HIV) infection.
5. History of allogeneic tissue/solid organ transplant.
6. History or clinical evidence of central nervous system (CNS) metastases without exceptions
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to LSTA1 or other agents used in the study, including those discovered by other ongoing studies of LSTA1 or other agents used in the study.
8. Existing venous thromboembolism at the time of CRS-HIPEC.
9. Severe or uncontrolled medical disorder that would, in the investigator's opinion, impair ability to undergo CRS-HIPEC and receive study treatment. This includes, but is not limited to the following laboratory values and other parameters within 30 days prior to planned date of CRS-HIPEC:

   1. Platelets < 100,000/mm3
   2. White blood cell count < 3000/ mm3
   3. Absolute neutrophil count < 1,500/mm3
   4. Serum albumin < 2.5 g/L
   5. Alanine transaminase (ALT) and aspartate aminotransferase (AST) > 2.5 x upper limit of normal (ULN) in the absence of liver metastases or > 5 x ULN in the presence of liver metastases
   6. Bilirubin > 1.5 x ULN
   7. Glomerular Filtration Rate (per Modification of Diet in Renal Disease equation) < 30 mL/min
   8. Hemoglobin < 9.0 g/dL (drawn 24 hours after a transfusion, if relevant)
   9. International normalised ratio (INR) > 2.0 (for patients not receiving therapeutic anticoagulation)
   10. Adequate respiratory and cardiac function (PaO2 ≥ 60 mm Hg or oxygen saturation ≥ 92% on room air, and 12-lead electrocardiogram (ECG) with normal tracing or QT interval < 470 ms)
10. Participants who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Adverse events of interest (AE-I) | postoperatively from the date of CRS-HIPEC to date of discharge (typically 1-2 weeks)
  The proportion of subjects experiencing an inpatient adverse event of interest (AE-I; gastrointestinal fistula/leak, neutropenia, intra-abdominal abscess, venous thromboembolism, mortality)
Drug concentration in tumor | at time of surgery
  Total drug content in tumor, divided by total tumor mass

SECONDARY OUTCOMES:
Progression-Free Survival and Overall Survival | 5 years
  Time (in months) from randomization to time of progression or death due to any cause, whichever occurs first (PFS), or to time of death due to any cause (OS).
Adverse Events (AEs) | 30 Days
  Incidence of any adverse events (AEs) by grade and system organ class using CTCAE v5.0 up to 30 days from the date of CRS-HIPEC.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Baumgartner, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States